CLINICAL TRIAL: NCT03644446
Title: Bisoprolol Plasma Residual Concentrations for the Optimization of Drug Management in Heart Failure With Mild to Reduced Ejection Fraction
Brief Title: Bisoprolol Plasma Residual Concentrations in Chronic Heart Failure
Acronym: PREVALENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: DC-2016-2725
Record Dates: First submitted 2018-08-13; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Bisoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — One blood sample for each patient at the time of inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bisoprolol 5mg: Chronic heart failure with mild to reduced ejection fraction adult patients with bisoprolol intakes at 5mg (patient's maximum tolerated dose), stable, with a left ventricular ejection fraction < 50%. Consecutive patients at the CHU de Caen.
  Interventions: Biological: Bisoprolol plasma residual concentration dosage
- Bisoprolol 7.5mg: Chronic heart failure with mild to reduced ejection fraction adult patients with bisoprolol intakes at 7.5mg (patient's maximum tolerated dose), stable, with a left ventricular ejection fraction < 50%. Consecutive patients at the CHU de Caen.
  Interventions: Biological: Bisoprolol plasma residual concentration dosage
- Bisoprolol 10mg: Chronic heart failure with mild to reduced ejection fraction adult patients with bisoprolol intakes at 10mg (patient's maximum tolerated dose), stable, with a left ventricular ejection fraction < 50%. Consecutive patients at the CHU de Caen.
  Interventions: Biological: Bisoprolol plasma residual concentration dosage

INTERVENTIONS:
Biological: Bisoprolol plasma residual concentration dosage — Bisoprolol plasma residual concentration dosage will be subsequently studied by renal function (altered if creatinine clearance < 30mL/min, mild altered between 30-60mL/min, normal > 60mL/min as estimated by the CKD-EPI formula)

SUMMARY:
This study evaluate the dosage of bisoprolol plasma residual concentrations in chronic heart failure with mild to reduced ejection fraction adult patients by dose and renal function.

DETAILED DESCRIPTION:
The clinical relevance of bisoprolol plasma residual concentration in the management of HF medical therapy and the impact of renal function on reaching the maximum tolerated dose has never been studied. The investigators will perform an observational study to answer this issue.

In this study, there will be no changes of the doses of bisoprolol, whatever the bisoprolol plasma concentration, with the exception of vital threatening concentrations. This study is a pilot study.

Participants will be consecutive ambulatory chronic heart failure patients followed at the CHU de Caen, treated with maximum tolerated dose of bisoprolol with mild to reduced ejection fraction. Participants can benefit of the other heart failure recommended treatment at the exception of ivabradine that would confound the bisoprolol effect on heart rate. Participants will be subsequently studied by renal function.

Patients will be followed at one year with the electronic health record of the CHU de Caen for clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive ambulatory patients with chronic heart failure with mild to reduced ejection fraction (LVEF < 50%) at the CHU de Caen
* Aged 18 y.o. or older
* With a stable heart failure (see exclusion criteria)
* At the maximum tolerated dose of bisoprolol for at least one week (maximum dose reached without adverse tolerance event: orthostatic hypotension, symptomatic bradycardia, fatigue related to the treatment)

Exclusion Criteria:

* Unstable HF, that are patients who presented in the last 3 months before inclusion an hospitalization for any cardiovascular event including HF, new onset or worsening of HF or coronary artery disease symptoms
* Patient refusing to participate
* Patients with a non maximum tolerated dose of bisoprolol
* Patients with ivabradine intakes
* Body weight < 60kg or > 100kg
* Severe liver insufficiency
* Pregnancy
* Liberty deprived patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive ambulatory chronic HFrEF patients followed at the CHU de Caen, treated with maximum tolerated dose of bisoprolol. Patients can benefit of other HFrEF recommended treatment at the exception of ivabradine that would confound the bisoprolol effect on heart rate. Patients will be subsequently studied by renal function (altered if creatinine clearance < 30mL/min, mild altered between 30-60mL/min, normal > 60mL/min as estimated by the CKD-EPI formula) and bisoprolol dose (5, 7.5 or 10mg).
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-11-02 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
Bisoprolol residual plasma concentration by dose and renal function | At the time of inclusion
  Bisoprolol plasma residual concentrations will be performed by liquid chromatography with tandem mass spectrometry (LC-MS/MS) with simple precipitation of proteins with acetonitrile, as described by Liu et al. The quantification will be in positive mode by multiple reaction monitoring with the following transitions: 326 to 116 for bisoprolol and 256 to 167 for diphenhydramine (control). Bisoprolol concentrations will be expressed in µg/L.

SECONDARY OUTCOMES:
Clinical parameters at the time of inclusion | At the time of inclusion
  Heart rate in beats per minute (bpm). Heart rate will be studied as a continous outcome and as a dichotomous outcome for efficacy. The efficacy parameter cutoff is a heart rate < 70bpm.
Clinical parameters at the time of inclusion | At the time of inclusion
  Systolic and diastolic blood pressure (in mmHg)
Clinical parameters at the time of inclusion | At the time of inclusion
  Tolerance : presence of any new symptom that requires a dose lowering or discontinuation of bisoprolol (dichotomous outcome) or symptomatic orthostatic hypotension
Clinical parameters at the time of inclusion | At the time of inclusion
  Tolerance : presence of a symptomatic orthostatic hypotension (dichotomous outcome) that is defined as a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg within three minutes of standing when compared with blood pressure from the sitting or supine position.
Biological assessment | At the time of inclusion
  Routine biological evaluation : creatinine (in µmol/L)
Biological assessment | At the time of inclusion
  Routine biological evaluation : Brain Natriuretic Peptide (in pg/mL)
Biological assessment | At the time of inclusion
  Galectin-3 (in ng/mL)
Clinical outcomes at one year | At one year follow-up
  Heart failure symptoms worsening (dichotomous variable)
Clinical outcomes at one year | At one year follow-up
  Hospitalization for heart failure (dichotomous variable)
Clinical outcomes at one year | At one year follow-up
  Death from any cause (dichotomous variable)
Clinical outcomes at one year | At one year follow-up
  Bisoprolol dose modification (categorical variable : dose increased, dose decreased, dose unchanged and quantitative analysis of mean change between bisoprolol inclusion dose and bisoprolol dose at one year).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurray JJ, Stewart S. Epidemiology, aetiology, and prognosis of heart failure. Heart. 2000 May;83(5):596-602. doi: 10.1136/heart.83.5.596. No abstract available. PMID 10768918
- [Background] Mosterd A, Hoes AW. Clinical epidemiology of heart failure. Heart. 2007 Sep;93(9):1137-46. doi: 10.1136/hrt.2003.025270. PMID 17699180
- [Background] Stewart S, MacIntyre K, Hole DJ, Capewell S, McMurray JJ. More 'malignant' than cancer? Five-year survival following a first admission for heart failure. Eur J Heart Fail. 2001 Jun;3(3):315-22. doi: 10.1016/s1388-9842(00)00141-0. PMID 11378002
- [Background] Stewart S, Ekman I, Ekman T, Oden A, Rosengren A. Population impact of heart failure and the most common forms of cancer: a study of 1 162 309 hospital cases in Sweden (1988 to 2004). Circ Cardiovasc Qual Outcomes. 2010 Nov;3(6):573-80. doi: 10.1161/CIRCOUTCOMES.110.957571. Epub 2010 Oct 5. PMID 20923990
- [Background] Jhund PS, Macintyre K, Simpson CR, Lewsey JD, Stewart S, Redpath A, Chalmers JW, Capewell S, McMurray JJ. Long-term trends in first hospitalization for heart failure and subsequent survival between 1986 and 2003: a population study of 5.1 million people. Circulation. 2009 Feb 3;119(4):515-23. doi: 10.1161/CIRCULATIONAHA.108.812172. Epub 2009 Jan 19. PMID 19153268
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522
- [Background] Bristow MR. Treatment of chronic heart failure with beta-adrenergic receptor antagonists: a convergence of receptor pharmacology and clinical cardiology. Circ Res. 2011 Oct 28;109(10):1176-94. doi: 10.1161/CIRCRESAHA.111.245092. PMID 22034480
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II): a randomised trial. Lancet. 1999 Jan 2;353(9146):9-13. PMID 10023943
- [Background] Effect of metoprolol CR/XL in chronic heart failure: Metoprolol CR/XL Randomised Intervention Trial in Congestive Heart Failure (MERIT-HF). Lancet. 1999 Jun 12;353(9169):2001-7. PMID 10376614
- [Background] Hjalmarson A, Goldstein S, Fagerberg B, Wedel H, Waagstein F, Kjekshus J, Wikstrand J, El Allaf D, Vitovec J, Aldershvile J, Halinen M, Dietz R, Neuhaus KL, Janosi A, Thorgeirsson G, Dunselman PH, Gullestad L, Kuch J, Herlitz J, Rickenbacher P, Ball S, Gottlieb S, Deedwania P. Effects of controlled-release metoprolol on total mortality, hospitalizations, and well-being in patients with heart failure: the Metoprolol CR/XL Randomized Intervention Trial in congestive heart failure (MERIT-HF). MERIT-HF Study Group. JAMA. 2000 Mar 8;283(10):1295-302. doi: 10.1001/jama.283.10.1295. PMID 10714728
- [Background] Packer M, Fowler MB, Roecker EB, Coats AJ, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Staiger C, Holcslaw TL, Amann-Zalan I, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival (COPERNICUS) Study Group. Effect of carvedilol on the morbidity of patients with severe chronic heart failure: results of the carvedilol prospective randomized cumulative survival (COPERNICUS) study. Circulation. 2002 Oct 22;106(17):2194-9. doi: 10.1161/01.cir.0000035653.72855.bf. PMID 12390947
- [Background] Pasternak B, Mattsson A, Svanstrom H, Hviid A. Comparative effectiveness of bisoprolol and metoprolol succinate in patients with heart failure. Int J Cardiol. 2015;190:4-6. doi: 10.1016/j.ijcard.2015.03.441. Epub 2015 Apr 18. No abstract available. PMID 25912106
- [Background] Fiuzat M, Wojdyla D, Kitzman D, Fleg J, Keteyian SJ, Kraus WE, Pina IL, Whellan D, O'Connor CM. Relationship of beta-blocker dose with outcomes in ambulatory heart failure patients with systolic dysfunction: results from the HF-ACTION (Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training) trial. J Am Coll Cardiol. 2012 Jul 17;60(3):208-15. doi: 10.1016/j.jacc.2012.03.023. Epub 2012 May 2. PMID 22560018
- [Background] Fiuzat M, Wojdyla D, Pina I, Adams K, Whellan D, O'Connor CM. Heart Rate or Beta-Blocker Dose? Association With Outcomes in Ambulatory Heart Failure Patients With Systolic Dysfunction: Results From the HF-ACTION Trial. JACC Heart Fail. 2016 Feb;4(2):109-115. doi: 10.1016/j.jchf.2015.09.002. Epub 2015 Oct 28. PMID 26519996
- [Background] Fonarow GC, Abraham WT, Albert NM, Stough WG, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB. Dosing of beta-blocker therapy before, during, and after hospitalization for heart failure (from Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure). Am J Cardiol. 2008 Dec 1;102(11):1524-9. doi: 10.1016/j.amjcard.2008.07.045. Epub 2008 Sep 6. PMID 19026308
- [Background] Dungen HD, Apostolovic S, Inkrot S, Tahirovic E, Krackhardt F, Pavlovic M, Putnikovic B, Lainscak M, Gelbrich G, Edelmann F, Wachter R, Eschenhagen T, Waagstein F, Follath F, Rauchhaus M, Haverkamp W, Osterziel KJ, Dietz R; CIBIS-ELD Investigators, Subproject Multicenter Trials in the Competence Network Heart Failure. Bisoprolol vs. carvedilol in elderly patients with heart failure: rationale and design of the CIBIS-ELD trial. Clin Res Cardiol. 2008 Sep;97(9):578-86. doi: 10.1007/s00392-008-0681-6. Epub 2008 Jun 9. PMID 18542839
- [Background] Gelbrich G, Edelmann F, Inkrot S, Lainscak M, Apostolovic S, Neskovic AN, Waagstein F, Loeffler M, Anker SD, Dietz R, Dungen HD; CIBIS-ELD investigators. Is target dose the treatment target? Uptitrating beta-blockers for heart failure in the elderly. Int J Cardiol. 2012 Feb 23;155(1):160-6. doi: 10.1016/j.ijcard.2011.11.018. Epub 2011 Nov 30. PMID 22133470
- [Background] Kirch W, Rose I, Demers HG, Leopold G, Pabst J, Ohnhaus EE. Pharmacokinetics of bisoprolol during repeated oral administration to healthy volunteers and patients with kidney or liver disease. Clin Pharmacokinet. 1987 Aug;13(2):110-7. doi: 10.2165/00003088-198713020-00003. PMID 2887325
- [Background] Fisher ML, Gottlieb SS, Plotnick GD, Greenberg NL, Patten RD, Bennett SK, Hamilton BP. Beneficial effects of metoprolol in heart failure associated with coronary artery disease: a randomized trial. J Am Coll Cardiol. 1994 Mar 15;23(4):943-50. doi: 10.1016/0735-1097(94)90641-6. PMID 8106700
- [Background] Olsen SL, Gilbert EM, Renlund DG, Taylor DO, Yanowitz FD, Bristow MR. Carvedilol improves left ventricular function and symptoms in chronic heart failure: a double-blind randomized study. J Am Coll Cardiol. 1995 May;25(6):1225-31. doi: 10.1016/0735-1097(95)00012-S. PMID 7722114
- [Background] Metra M, Nardi M, Giubbini R, Dei Cas L. Effects of short- and long-term carvedilol administration on rest and exercise hemodynamic variables, exercise capacity and clinical conditions in patients with idiopathic dilated cardiomyopathy. J Am Coll Cardiol. 1994 Dec;24(7):1678-87. doi: 10.1016/0735-1097(94)90174-0. PMID 7963115
- [Background] Krum H, Sackner-Bernstein JD, Goldsmith RL, Kukin ML, Schwartz B, Penn J, Medina N, Yushak M, Horn E, Katz SD, et al. Double-blind, placebo-controlled study of the long-term efficacy of carvedilol in patients with severe chronic heart failure. Circulation. 1995 Sep 15;92(6):1499-506. doi: 10.1161/01.cir.92.6.1499. PMID 7664433
- [Background] Packer M, Coats AJ, Fowler MB, Katus HA, Krum H, Mohacsi P, Rouleau JL, Tendera M, Castaigne A, Roecker EB, Schultz MK, DeMets DL; Carvedilol Prospective Randomized Cumulative Survival Study Group. Effect of carvedilol on survival in severe chronic heart failure. N Engl J Med. 2001 May 31;344(22):1651-8. doi: 10.1056/NEJM200105313442201. PMID 11386263
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Randomised, placebo-controlled trial of carvedilol in patients with congestive heart failure due to ischaemic heart disease. Australia/New Zealand Heart Failure Research Collaborative Group. Lancet. 1997 Feb 8;349(9049):375-80. PMID 9033462
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology; Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S, McDonagh T, Sechtem U, Bonet LA, Avraamides P, Ben Lamin HA, Brignole M, Coca A, Cowburn P, Dargie H, Elliott P, Flachskampf FA, Guida GF, Hardman S, Iung B, Merkely B, Mueller C, Nanas JN, Nielsen OW, Orn S, Parissis JT, Ponikowski P; ESC Committee for Practice Guidelines. ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2012 Aug;14(8):803-69. doi: 10.1093/eurjhf/hfs105. No abstract available. PMID 22828712
- [Background] Liu M, Zhang D, Sun Y, Wang Y, Liu Z, Gu J. Liquid chromatographic-electrospray tandem mass spectrometric determination of bisoprolol in human plasma. Biomed Chromatogr. 2007 May;21(5):508-13. doi: 10.1002/bmc.785. PMID 17294507